CLINICAL TRIAL: NCT06074692
Title: A Prospective Phase II Study of PARP Inhibition and Check Point-inhibition Immunotherapy With Concurrent Stereotactic Body Radiotherapy (SBRT) in Patients With Metastatic or Advanced Sarcoma
Brief Title: PARP Inhibition, Stereotactic Body Radiotherapy and Immunotherapy for Metastatic or Advanced Sarcoma (PRIMA)
Acronym: PRIMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Weibin Zhang, MD, PhD., Chief director of the orthopaedics department, Vice director of the orthpaedic research institute of Shanghai Jiaotong University, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-LLS-220
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Sarcoma; Sarcoma,Soft Tissue; Sarcoma of Bone
Keywords: sarcoma; bone and soft tissue sarcoma; PARP inhibitor; SBRT; checkpoint inhibitor
MeSH Terms: conditions — Sarcoma; Osteosarcoma | interventions — camrelizumab; fluzoparib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bone arm (Experimental): Bone tumor subgroup (bone arm) includes high-grade osteosarcoma, chondrosarcoma, undifferentiated bone sarcoma and other rare bone sarcomas with complex genomic features..
  Interventions: Combination Product: Camrelizumab and fluzoparib with concurrent stereotactic body radiotherapy (SBRT)
- Soft tissue arm (Experimental): Soft tissue sarcoma subgroup (soft tissue arm) includes leiomyosarcoma, pleomorphic rhabdomyosarcoma, angiosarcoma, fibrosarcoma, epithelioid sarcoma, malignant peripheral nerve sheath tumor(MPNST) and other rare soft tissue sarcomas with complex genomic features.
  Interventions: Combination Product: Camrelizumab and fluzoparib with concurrent stereotactic body radiotherapy (SBRT)
- UPS/DDLPS arm (Experimental): Immune hot tumor subgroup (UPS/DDLPS arm) includes undifferentiated pleomorphic sarcoma (UPS), dedifferentiated liposarcoma (DDLPS).
  Interventions: Combination Product: Camrelizumab and fluzoparib with concurrent stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Combination Product: Camrelizumab and fluzoparib with concurrent stereotactic body radiotherapy (SBRT) — Patients receive Camrelizumab (PD-1 inhibitor) and fluzoparib (PARP inhibitor) with concurrent stereotactic body radiotherapy (SBRT)

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of PARP Inhibition and programmed cell death protein-1 (PD-1) blockade immunotherapy with concurrent stereotactic body radiotherapy (SBRT) for metastatic or advanced bone and soft tissue sarcoma.

DETAILED DESCRIPTION:
Bone and soft tissue sarcomas are a group of highly heterogeneous malignant tumors that originate from mesenchymal tissue. The recurrent and metastatic sarcomas are usually refractory to traditional radiotherapy and chemotherapy, with a five-year survival rate is less than 20% to 30%. Therefore, novel therapy targeting the molecular phenotypic characteristics of bone and soft tissue sarcomas and conduct personalized and precise treatment for specific target patient subgroups is one of the important directions in the current clinical and translational fields.

Studies based on the anti-cancer mechanism of synthetic lethality have shown that tumor cells with BRCA1 or BRCA2 gene mutations are very sensitive to the action of PARP inhibitors. Interestingly, recent research results have shown that many other tumor types besides gynecological tumors can also exhibit BRCA-like phenotypes (BRCAness) and genomic instability (GI). Among them, BRCAness is a subtype of bone and soft tissue sarcoma with poor prognosis. Although such patients rarely carry BRCA gene mutations, they can still potentially benefit from treatment with drugs related to DNA damage and synthetic lethality, such as PARP inhibitors. In addition, the latest research shows that the BRCA-like phenotype in sarcoma is related to immunosuppression in its tumor microenvironment and targeted intervention of the PARP pathway is likely to have a potential immune sensitizing effect on the tumor microenvironment of sarcoma. Our previous study based on 264 samples also suggested that in sarcoma subtypes with genomic complexity, tumor cells often demonstrated high GI characteristics, and the corresponding tumor transcriptomes exhibited BRCAness. Furthermore, the investigators established 8 cases of patient-derived sarcoma primary cell model (PTCC) through tumor biopsy samples and observed a high sensitivity to DNA damage in sarcoma habouring BRCAness.

In recent years, studies have found that when radiotherapy is given to local tumor lesions, Abscopal effect could be elicited by the immunogenic death of the local tumor. The investigators recently reviewed the clinical prognosis of 44 patients with advanced bone and soft tissue sarcoma treated with stereotactic body radiation therapy (SBRT) in our institute and found that the tumor response rate to the immune checkpoint inhibitor appears to be significantly increased after SBRT. Based on these findings, the investigators speculate that the combination of SBRT and PARP inhibition regimens could potentially boost the immunogenic death and further improve the immunotherapy response in metastatic or advanced sarcomas.

In this clinical trial, the investigators aim to evaluate the efficacy and safety of PARP Inhibition and programmed cell death protein-1 (PD-1) blockade immunotherapy with concurrent stereotactic body radiotherapy (SBRT) for metastatic or advanced bone and soft tissue sarcoma as a phase II clinical study. Meanwhile, the investigators evaluated the patient's tumor gene mutation, homologous recombination deficiency (HRD) score, and RAD51 functional testing and other aspects for correlative biomarker exploration, providing a theoretical basis for molecular precision treatment of bone and soft tissue sarcoma with PARP inhibitiors.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed before any trial-related procedures are carried out
2. Histologically confirmed high-grade sarcoma of bone or soft tissue; the lesion has distant metastasis or is locally advanced and cannot be completely resected at the time of enrollment, or the patient cannot tolerate or refuses surgical resection;
3. Have received at least one systemic treatment regimen(s) at the time of enrollment, and have not received prior PARP inhibitor treatment.
4. With measurable lesions according to Response Evaluation Criteria in Solid Tumors (RECIST1.1);
5. Aged no less than 10 years old and no more than 70 years old;
6. For patients ≥16 years old, ECOG score is between 0 and 2 (for patients with amputations, if they can basically take care of themselves and can move freely for more than 50% of their waking hours with the assistance of stretchers, walkers, wheelchairs, etc.) still included);
7. For patients under 16 years old, Lansky score is at least 70 or above (for patients with amputations who are unable to participate in active recreational activities due to amputation), if they can participate in most active recreational activities with the assistance of walkers, wheelchairs, etc., they are still eligible included).
8. The expected survival time is greater than 24 weeks;
9. The majority of the recurrent lesions with an established radiological diagnosis could receive SBRT;
10. Major organ functions meet basic safety standards within 7-14 days before treatment.
11. Women of childbearing age should agree that they must use contraceptive measures (such as intrauterine devices, birth control pills or condoms) during the study and within 6 months after the end of the study; if in doubt, serum or urine tests within 7 days before study enrollment The pregnancy test is negative and the patient must be non-lactating; the male should agree that contraceptive measures must be used during the study period and within 6 months after the end of the study period;
12. If there are recurrent lesions previously treated by surgery, radiofrequency ablation or radiotherapy:

    1. If the image of the metastatic lesion is stable, enrollment is allowed and SBRT is not required for that lesion;
    2. If the metastatic lesion has image progression, if it was previously treated with surgery and SBRT can be performed, enrollment is allowed; if it was previously treated with radiofrequency ablation or radiotherapy, if repeat SBRT can be considered, enrollment is allowed.

Exclusion Criteria:

1. Diagnosed with malignant diseases other than tumors within 5 years before the first dose;
2. Currently participating in interventional clinical research treatment, or have received other research drugs or used research equipment within 4 weeks before the first dose;
3. Previously received the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs targeting another stimulating or synergistic inhibition of T cell receptors (e.g., CTLA-4, OX-40, CD137) drug and secondary resistance to the drug (i.e., the best efficacy evaluation is CR, PR or SD lasting more than 4 months, but secondary tumor resistance develops after treatment).
4. Received systemic systemic treatment with Chinese patent medicines with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except local use to control pleural effusion) within 2 weeks before the first dose;
5. Active autoimmune disease requiring systemic treatment (such as use of disease-modifying drugs, glucocorticoids, or immunosuppressants) within 2 years before the first dose. Replacement therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatments;
6. Are receiving systemic glucocorticoid treatment (excluding nasal spray, inhaled or other route of topical glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first dose of the study;
7. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
8. Known to be allergic to any components of monoclonal antibody preparations (have experienced grade 3 or above allergic reactions);
9. Have not fully recovered from toxicity and/or complications caused by any intervention before initiating treatment (i.e., ≤Grade 1 or reaching baseline, excluding fatigue or alopecia);
10. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV1/2 antibody positive);
11. Get live vaccine within 30 days before the first dose (cycle 1, day 1);
12. Pregnant or lactating women;
13. Any serious or uncontrollable systemic disease

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
6-momth progression-free survival rate (6m-PFSR) | 6 months from recruitment
  The proportion of patients that are progression-free according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), defined as the ratio of patients who have not died or progressed (CR+PR+SD) over the total number of subjects recruited.

SECONDARY OUTCOMES:
Objective respones rate (ORR) | From baseline to disease progression or death, whichever occurs first, until 3 years after accrual
  Defined as the number of subjects with a best response of (CR+PR)/total number of subjects*100% based on RECISTv1.1 and irRECIST standards respectively
Disease control rate (DCR) | From baseline to disease progression or death, whichever occurs first, up to 3 years after accrual
  Defined as the number of subjects with a best response of (CR+PR+SD)/total number of subjects*100% based on RECISTv1.1 and irRECIST standards respectively;
Duration of response (DOR) | From baseline to disease progression or death, whichever occurs first, up to 3 years after accrual
  Defined as the interval from first time of response (CR or PR) until disease progression (PD) according to RECISTv1.1 and irRECIST standards respectively, and estimated by the Kaplan-Meier method, including median, Interquartiles and 95% confidence intervals
Progression-free survival (PFS) | From baseline to disease progression or death, whichever occurs first, up to 3 years after accrual
  Defined as the time from receiving the first study drug to the death or relapse of the subject, assessed by RECISTv1.1 and irRECIST standards respectively, and estimated by the Kaplan-Meier method, including median, quartile and 95% confidence interval
Overall survival (OS) | From baseline until the reported death of the patients due to any causes, up to 3 years after accrual
  defined as the time from receiving the first study drug treatment to the subject's death, estimated by the Kaplan-Meier method, including median, quartile and 95% confidence interval;
Quality of life assessed by patient-reported outcomes (PROs) | From baseline until the reported death of the patients due to any causes, up to 3 years after accrual
  The quality of life score using PROs based on EORTC QLQ-C30 scale (adult) or Paediatric Quality of Life Inventory (PedsQL) scale at baseline and at each followed up after treatment.
Number of participants with adverse events | From the first dose of study treatment to 30 days after the last dose of study treatment or before the start day of new anti-cancer drug therapy, whichever occurs first, up to 3 years.
  Number of participants with Treatment emergent adverse events (TEAE) and serious adverse events (SAE). AE was defines as any toxicities in a participant who received study therapy irrespective of the causal relationship. SAE was defined as one of the following: was fatal or life-threatening; resulted in persistent or significant disability/incapacity or inpatient hospitalization or prolongation of existing hospitalization.

OTHER OUTCOMES:
Exploratory outcome: progression-free survival(PFS) in different subgroup | From baseline to disease progression or death, whichever occurs first, up to 3 years after accrual.
  The PFS for each subgroups in terms of clinicopathological and genomic characteristics (age, gender, histological type, solitary or multiple metastases, unilateral or bilateral metastases, early or late metastases, calcifying or non-calcifying lesions, with or without lesion cavitation, with or without AEs, etc.
Exploratory outcome: the homologous recombination deficiency (HRD) score in tumor samples | From baseline to disease progression or death, whichever occurs first, up to 3 years after accrual
  The correlative relationship between the tumor response and the genomic biomarker (i.e.
  homologous recombination-related [HRR] gene mutation, homologous recombination deficiency (HRD) score (LOH+TAI+LST), and RAD51 functional testing) and the therapeutic outcome.
Exploratory outcome: the expression of immune infiltration biomarker in tumor samples | From baseline to disease progression or death, whichever occurs first, up to 3 years after accrual.
  Tumor microenvironment change (immune infiltration, PD-1/PD-L1 expression, immunogenic death, etc.) pre- and post- SBRT, and conduct correlative analysis between these immune microenvironment indeces and the therapeutic outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Weibin Zhang, PhD, MD, Principal Investigator — Ruijin Hospital; Yuhui Shen, PhD, MD, Principal Investigator — Ruijin Hospital; Qiyuan Bao, PhD, MD, Principal Investigator — Ruijin Hospital; Junxiang Wen, PhD, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
individual participant data (IPD) will be available to academic research upon reasonable request, under the local offical rules and regulations.